CLINICAL TRIAL: NCT03119389
Title: Efficacy of a Direct Gloving Strategy to Improve Compliance With Infection Prevention Practices: A Cluster-randomized Trial
Brief Title: Direct Gloving Strategy: A Cluster-randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kerri A Thom, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00065259
Record Dates: First submitted 2017-03-30; First posted 2017-04-18 (Actual); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Hand Hygiene
Keywords: Hand Hygiene; Non-sterile glove use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donning Non-Sterile Gloves without HH (Experimental): In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves is NOT necessary. For Aim A, observations will be made on compliance at entry and exit with hand hygiene and glove use. For Aim B, samples will be obtained from the gloves after donning to determine total aerobic colony counts and to identify important hospital pathogens
  Interventions: Behavioral: Donning Non-Sterile Gloves without HH
- HH before donning Non-Sterile Gloves (No Intervention): In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves IS necessary. For Aim A, observations will be made on compliance at entry and exit with hand hygiene and glove use. For Aim B, samples will be obtained from the gloves after donning to determine total aerobic colony counts and to identify important hospital pathogens

INTERVENTIONS:
Behavioral: Donning Non-Sterile Gloves without HH — Current practice is to perform hand hygiene before donning of non-sterile gloves. In units assigned to the intervention, healthcare workers within the units will be educated that performing hand hygiene before donning non-sterile gloves is not necessary.
  Arms: Donning Non-Sterile Gloves without HH

SUMMARY:
The necessity of Hand hygiene (HH) before donning non-sterile gloves is unknown. Furthermore, because of the additional time required to cleanse hands and then don gloves, as well as the cumbersome nature of applying gloves to recently washed hands, this practice leads to non-compliance with both HH and glove use - placing patients at risk. In a pilot study, the investigators performed a randomized trial of 230 healthcare workers and demonstrated no difference in total bacterial colony counts or identification of pathogenic bacteria from the gloves of persons who either performed HH or did not perform HH prior to putting on non-sterile gloves. If unnecessary, HH before non-sterile glove use wastes valuable time, which might otherwise be spent engaged in direct patient care. And removing this unnecessary step may lead to increased compliance with infection prevention measures. In Aim A, the investigators will perform a multi-center randomized control trial to evaluate the efficacy of a direct gloving strategy to improve compliance with infection prevention practices. In Aim B, the investigators will perform a nested multi-center validation study, where the gloved hands of healthcare workers will be randomly sampled to determine bacterial contamination of non-sterile gloves after donning.

DETAILED DESCRIPTION:
This study seeks to investigate alternative strategies to hand hygiene (HH) and glove use in situations where glove use is required to perform health care activities in an effort to increase compliance with infection prevention efforts.

HH is the cornerstone of infection prevention. Despite the importance of and increased focus on HH, compliance remains low in healthcare settings (40% on average in a large meta-analysis). Insufficient time, high workload and under staffing are important barriers. Glove use, which is common and increasing, is another major barrier. New strategies are needed that improve time and efficiency particularly in settings where glove use is required (e.g. Contact Precautions). One area for further study is the requirement for HH prior to non-sterile glove use. This is a recommended practice with poor compliance that may be unnecessary. Furthermore, it may lead to reduced compliance with other recommended infection prevention practices, such as glove use. In this proposal the investigators identify a novel strategy of directly gloving without performing HH prior to non-sterile glove use as a potential solution.

In this study the investigators aim to perform a multicenter, cluster-randomized trial to evaluate the efficacy of direct gloving to improve compliance with infection prevention practices (i.e. HH and glove use). Herein, the investigators will evaluate the safety and efficacy of directly gloving (compared to performing HH prior to glove use) and assess whether this strategy will lead to increased compliance with both HH and glove use. The investigators previously demonstrated the safety of this strategy in a single-center randomized controlled pilot trial where the investigators found no difference in bacterial contamination of gloves of healthcare providers who either performed or did not perform HH prior to donning non-sterile gloves. Thus, with potentially no added benefit and in a setting where the investigators know that HH compliance is the lowest (i.e. prior to glove use), mandating HH prior to donning gloves as recommended in current guidelines could actually reduce both HH and glove compliance, placing patients at increased risk for developing infection.

ELIGIBILITY:
For Aim B

Inclusion Criteria:

* Health professional at one of the study sites
* Has direct interaction with patients at study sites (healthcare worker)

Exclusion Criteria:

* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14418 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Thom, MD, MS, Principal Investigator — University of Maryland, College Park
Locations (3):
- United States (3):
  - University of Iowa Hospitals, Iowa City, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thom KA, Rock C, Robinson GL, Reisinger HS, Baloh J, Li S, Diekema DJ, Herwaldt LA, Johnson JK, Harris AD, Perencevich EN. Direct Gloving vs Hand Hygiene Before Donning Gloves in Adherence to Hospital Infection Control Practices: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2336758. doi: 10.1001/jamanetworkopen.2023.36758. PMID 37883088

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Units within each hospital were recruited to participate in the baseline study. Observation of healthcare worker hand hygiene and glove use were observed during the baseline period. Units with similar hand hygiene and glove use compliance were approached for participation in the study.
Units Other Than Participants: healthcare units
Groups:
- HH Before Donning Non-Sterile Gloves: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves IS necessary. Individual healthcare workers within each unit were observed for the primary and secondary outcomes in order to obtain percentages for each outcome.
- Donning Non-Sterile Gloves Without HH: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves is NOT necessary.
  Donning Non-Sterile Gloves without HH: Current practice is to perform hand hygiene before donning of non-sterile gloves. In units assigned to the intervention, healthcare workers within the units will be educated that performing hand hygiene before donning non-sterile gloves is not necessary.
  Individual healthcare workers within each unit were observed for the primary and secondary outcomes in order to obtain percentages for each outcome.
Period: Overall Study
Arm/Group | HH Before Donning Non-Sterile Gloves | Donning Non-Sterile Gloves Without HH
Started | 6791; 7 healthcare units | 7627; 6 healthcare units
Completed | 6791; 7 healthcare units | 7627; 6 healthcare units
Not Completed | 0; 0 healthcare units | 0; 0 healthcare units

BASELINE CHARACTERISTICS:
Population: Healthcare workers are expected to perform hand hygiene before donning gloves when entering contact precaution rooms. In the baseline, healthcare worker compliance to performing hand hygiene before donning gloves was observed within each healthcare unit.
Units Other Than Participants: healthcare units
Groups:
- Donning Non-Sterile Gloves Without HH: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves is NOT necessary.
  Donning Non-Sterile Gloves without hand hygiene: Current practice is to perform hand hygiene before donning of non-sterile gloves. In units assigned to the intervention, healthcare workers within the units will be educated that performing hand hygiene before donning non-sterile gloves is not necessary.
  Individual healthcare workers within each unit were observed for the primary and secondary outcomes in order to obtain adherence to expected practice at entry to contact precaution rooms.
- HH Before Donning Non-Sterile Gloves: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves IS necessary.
  Individual healthcare workers within each unit were observed for the primary and secondary outcomes in order to obtain adherence to expected practice at entry to contact precaution rooms.
- Total: Total of all reporting groups
Arm/Group | Donning Non-Sterile Gloves Without HH | HH Before Donning Non-Sterile Gloves | Total
Number analyzed (Participants) | 633 | 927 | 1560
Number analyzed (healthcare units) | 6 | 7 | 13
Age, Customized [Count of Participants; unit: Participants]
  Unknown | 633 | 927 | 1560
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 633 | 927 | 1560
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Adherence to expected practice at entry to contact precaution rooms [Count of Participants; unit: Participants] | 236 | 282 | 518

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Compliance With Expected Infection Prevention Practices Upon Entry to Contact Precaution-patient Rooms
Description: Healthcare workers in the usual care group will be recorded as compliant if hand hygiene AND glove use is observed at room entry; healthcare workers in the intervention group only need to have glove use observed to be considered compliant.
Time Frame: 1 year
Population: The number analyzed is the number of observations made within each group of units randomized
Measure: Count of Participants; unit: Participants
Groups:
- Donning Non-Sterile Gloves Without Hand Hygiene: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves is NOT necessary.
  Donning Non-Sterile Gloves without hand hygiene: Current practice is to perform hand hygiene before donning of non-sterile gloves. In units assigned to the intervention, healthcare workers within the units will be educated that performing hand hygiene before donning non-sterile gloves is not necessary.
  Individual healthcare workers within each unit were observed for the primary outcome in order to obtain unit adherence for the primary outcome
- Hand Hygiene Before Donning Non-Sterile Gloves: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves IS necessary.
  Individual healthcare workers within each unit were observed for the primary outcome in order to obtain unit adherence for the primary outcome
Arm/Group | Donning Non-Sterile Gloves Without Hand Hygiene | Hand Hygiene Before Donning Non-Sterile Gloves
Number analyzed (Participants) | 1491 | 2299
Participants | 1297 | 954

2. Secondary Outcome: Proportion of Healthcare Worker Who Use Glove on Entry Into Contact Precaution Rooms
Description: Proportion of healthcare worker compliance with glove use upon entry to Contact Precaution-patient rooms for both groups
Time Frame: 1 year
Population: The number analyzed is the number of observations made within each group of units randomized
Measure: Count of Participants; unit: Participants
Groups:
- Donning Non-Sterile Gloves Without Hand Hygiene: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves is NOT necessary.
  Donning Non-Sterile Gloves without hand hygiene: Current practice is to perform hand hygiene before donning of non-sterile gloves. In units assigned to the intervention, healthcare workers within the units will be educated that performing hand hygiene before donning non-sterile gloves is not necessary.
- Hand Hygiene Before Donning Non-Sterile Gloves: In this arm, entire units will be assigned education that hand hygiene before donning non-sterile gloves IS necessary.
Arm/Group | Donning Non-Sterile Gloves Without Hand Hygiene | Hand Hygiene Before Donning Non-Sterile Gloves
Number analyzed (Participants) | 1491 | 2299
Participants | 1297 | 1530

3. Secondary Outcome: Proportion of Healthcare Workers Who Perform Hand Hygiene on Entry Into Non-contact Precaution Room
Description: Proportion of healthcare worker compliance with hand hygiene upon entry into non-contact precaution patient rooms
Time Frame: 1 year
Population: The number analyzed is the number of observations made within each group of units randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Donning Non-Sterile Gloves Without Hand Hygiene | Hand Hygiene Before Donning Non-Sterile Gloves
Number analyzed (Participants) | 1688 | 1315
Participants | 1111 | 951

4. Secondary Outcome: Proportion of Healthcare Worker Who Perform Hand Hygiene on Exit From Any Room
Description: Proportion of healthcare worker compliance with hand hygiene upon exit from any patient room
Time Frame: 1 year
Population: The number analyzed is the number of observations made within each group of units randomized
Measure: Count of Participants; unit: Participants
Arm/Group | Donning Non-Sterile Gloves Without Hand Hygiene | Hand Hygiene Before Donning Non-Sterile Gloves
Number analyzed (Participants) | 1785 | 1897
Participants | 1525 | 1587

5. Other Pre Specified Outcome: Mean Total Bacterial Colony Count
Description: Mean bacterial colony count from gloves of healthcare workers in the intervention and control units
Time Frame: 1 year
Population: The number analyzed is the number of observations made within each group of units randomized
Measure: Mean (Full Range); unit: Colony forming units
Arm/Group | Donning Non-Sterile Gloves Without Hand Hygiene | Hand Hygiene Before Donning Non-Sterile Gloves
Number analyzed (Participants) | 1194 | 1189
Colony forming units | 16.3 [0 to 300] | 9.5 [0 to 300]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the baseline of 6 months and intervention period of 1 year
Arm/Group | HH Before Donning Non-Sterile Gloves | Donning Non-Sterile Gloves Without HH
All-Cause Mortality (participants affected / at risk) | 0/6700 | 0/6158
Serious Adverse Events (participants affected / at risk) | 0/6700 | 0/6158
Other Adverse Events (participants affected / at risk) | 0/6700 | 0/6158

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-13): https://cdn.clinicaltrials.gov/large-docs/89/NCT03119389/Prot_SAP_000.pdf